CLINICAL TRIAL: NCT00379782
Title: Kukui Ahi Navigator Cancer Screening and Treatment Demonstration Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Responsible Party: Clayton Chong MD, Debbie Wong RN, Queen's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RA-2006-025
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer; Cervical Cancer; Prostate Cancer; Colorectal Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Lung Neoplasms

INTERVENTIONS:
Other: Navigation — Navigation and escourt

SUMMARY:
This Cancer Prevention and Treatment Demonstration Project funded by the Centers of Medicare and Medicaid Services awarded six sites across the United States to develop Patient Navigator Programs to eliminate disparities in the rate of preventative cancer screening and timely diagnosis and treatment of cancer for racial and ethnic minorities. This site of Molokai General Hospital are focused on Pacific Islanders and Asian Americans. This program called Kukui Ahi propose to increase screening and early detection for four targeted cancers-breast, cervical, colorectal, and prostate- with lung cancer additionally being included in treatment protocols to improve outcomes and satisfaction by employing a culturally appropriate navigation protocol to facilitate utilization of healthcare services and decrease health barriers.

The specific aims of the project is to:

1. Determine if a Navigator Program can reduce the proportion of the targeted cancers diagnosed at a late stage,
2. Determine if the Navigator Program can improve the continuity of health care for cancer patients,
3. Determine if the Navigator Program can improve quality of life and subjective well being of navigated cancer patients,
4. Determine if the Navigator Program is a cost-effective way to reduce cancer care disparities for screenable cancers.

DETAILED DESCRIPTION:
To be eligible, patients must have Medicare parts A and B, not enrolled in a managed care plan, not enrolled in hospice, and if currently have cancer, it must be either breast, cervical, colorectal, lung, or prostate. Patients may be enrolled up to 3 ½ years. After informed consent is obtained, the navigator will administer a CSA triage (attached) to determine if patient has cancer or not. Patients who have never had cancer or been in remission for five years are eligible for the screening arm and then will have the Screening CSA (attached) performed. Cancer screening arm of the study will then go into randomization.

Medistat has created a data entry system for randomization via internet. Medstat will create site administrators and CMS staff users. All users have a defined role that controls what they can see and do. Site administrators can perform all functions and create site staff users. Site staff users can only assign protocols. All users must supply a user identification and password to gain access to the site. Patients are qualified for the demonstration by site staff. Cancer status is ascertained via CSA. Sites will assign patient identification number that will be entered along with cancer status onto the website, no personal identification. RTI will then perform randomization protocol determination and log into database. Site reports available by sight only include individual protocol assignments by patient identification number, summarized protocol assignments by site and year, and view all individual assignments made within a time window. Only the site administrator can disenroll patients. RTI will be utilizing block randomization by site and arm (screening/treatment) in even blocks of 10-18 events depending on size of site.

The patients that are in the screening intervention group will have the navigational services. The control group will receive only nutritional education. Those patients who have non-study cancers and are not in remission for five years are ineligible for the study. The study cancers will be given a treatment CSA (attached). For those patients with study cancer, the patients will automatically be put in the navigational group. Molokai being such a small community where everyone knows everyone, it was agreed that to have a control group here would appear to be withholding care and cause bias. The control group will come from another community of similar demographics of Kahuku. Both navigational groups will have an initial CSA, annual CSA, and then an exit CSA conducted in the last six months of the program. CMS has not issued the annual or exit CSA at this time. Molokai has agreed to provide no more than 578 patients with delivery of navigational services to no more than 289 patients in the screening arm of the project.

Randomization to intervention or control group will be done as above per RTI International, a statistical firm contracted by CMS. Twenty-five cancer or treatment patients will be enrolled for navigational arm on Molokai and 25 control group patients from a neighboring island.

ELIGIBILITY:
Inclusion Criteria: Medicare Part A & B beneficiaries -

Exclusion Criteria: No medicare managed care or hospice beneficiaries, no other cancers other than target within 5 years remission.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 628 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
subject satisfaction with navigation | 7/2010

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Chong, MD, Principal Investigator — Molokai General Hospital/Queen's Medical Center
Locations (1):
- Molokai General Hospital, Kaunakakai, Hawaii, United States